CLINICAL TRIAL: NCT05744310
Title: Effects of Long Term Ventilation Support on the Quality of Life of ALS Patients and Their Families
Acronym: ALS-LTMV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Oslo University Hospital (Other); University Hospital, Akershus (Other); Helse Stavanger HF (Other Government); University Hospital of North Norway (Other); St. Olavs Hospital (Other); Nordland Hospital, Bodø (Unknown); Hospital of Southern Norway Kristiansand (Unknown); Østfold Hospital Kalnes (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 492102
Record Dates: First submitted 2023-01-30; First posted 2023-02-27 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2024-10

CONDITIONS: Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Nervous System Diseases; Spinal Cord Diseases; Neurodegenerative Diseases; TDP-43 Proteinopathies
Keywords: Quality of life; Overall quality of life; Health related quality of life; Disease specific quality of life; Ventilation support; Non-invasive ventilation support; Invasive ventilation support
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Nervous System Diseases; Spinal Cord Diseases; Neurodegenerative Diseases; TDP-43 Proteinopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ALS patients that choose life prolonging treatment with LTMV and their families (Active Comparator)
  Interventions: Device: Long term mechanical ventilation support
- ALS patients that decline life prolonging treatment with LTMV and their families (Active Comparator)
  Interventions: Device: No long term mechanical ventilation support

INTERVENTIONS:
Device: Long term mechanical ventilation support — Patients that choose life prolonging treatment with long term mechanical ventilation support
  Arms: ALS patients that choose life prolonging treatment with LTMV and their families
Device: No long term mechanical ventilation support — Patients that decline life prolonging treatment with long term mechanical ventilation support
  Arms: ALS patients that decline life prolonging treatment with LTMV and their families

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a serious rapidly progressive disease of the nervous system. The average survival from the time of diagnosis is two to three years. The patient physical and psychological sufferings in ALS are immense, and apart from Riluzole, there is no effective treatment. Care of advanced ALS have an estimated cost of 4-8 million NOK per year. Perhaps the most challenging topic of ALS care is the decision to extend ventilation support into the stages of disease that require treatment both during day and night. In these cases, treatment is clearly life-sustaining and although quality of life may be maintained, the burden of caregiving imposed upon family or health care workers is huge, regardless of tracheostomy (TIV) or non-invasive (NIV) modality.

The present study is a longitudinal questionnaire study in Norway measuring overall quality of life, health-related quality of life, and disease-specific quality of life in ALS patients, partners and children before and after the introduction of life sustaining ventilation support. The investigators aim to increase the knowledge on how life-sustaining ventilation support with NIV or TIV affects the quality of life in ALS patients, life partners and children. The results from the study may provide crucial information for clinicians and patients on one of the most difficult ethical issues of ALS treatment. The investigators anticipate that this information will facilitate a shared decision making processes, weighing benefits and disadvantages in a wider perspective.

ELIGIBILITY:
Inclusion criteria for patients:

1. A clinical diagnosis of probable ALS according to the revised El Escorial criteria
2. Progression of the illness leading the consulting physician to offer treatment with LTMV
3. Can communicate in Norwegian

Inclusion criteria for partners of ALS patients:

1. Partner of a patient with ALS with progression of the illness leading the consulting physician to offer treatment with LTMV
2. Can communicate in Norwegian

Inclusion criteria for children:

1. Children from 8 years and older having a parent who suffers from ALS with progression of the illness leading the consulting physician to offer treatment with LTMV
2. Can communicate in Norwegian

Exclusion criteria for patients, partners and children of ALS patients:

1. Potential participants with cognitive impairment or dementia.

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2032-08-21 (Estimated); Study Completion 2032-08-21 (Estimated)

PRIMARY OUTCOMES:
Overall quality of life assessed by the "Quality of Life Scale" | At inclusion
  "Quality of Life Scale" total score (range 16-112). Higher score indicates better quality of life.
Overall quality of life assessed by the "Quality of Life Scale" | 3 months after inclusion
  "Quality of Life Scale" total score (range 16-112). Higher score indicates better quality of life.
Overall quality of life assessed by the "Quality of Life Scale" | 9 months after inclusion
  "Quality of Life Scale" total score (range 16-112). Higher score indicates better quality of life.
Overall quality of life assessed by the "Quality of Life Scale" | 15 months after inclusion
  "Quality of Life Scale" total score (range 16-112). Higher score indicates better quality of life.
Overall quality of life assessed by the "Quality of Life Scale" | 21 months after inclusion
  "Quality of Life Scale" total score (range 16-112). Higher score indicates better quality of life.

SECONDARY OUTCOMES:
Health-related quality of life assessed by the "EQ-5D-5L" | At inclusion
  "EQ-5D-5L" index score and EQ-VAS score (range 0-100) where higher scores indicates better health-related quality of life.
Health-related quality of life assessed by the "EQ-5D-5L" | 3 months after inclusion
  "EQ-5D-5L" index score and EQ-VAS score (range 0-100) where higher scores indicates better health-related quality of life.
Health-related quality of life assessed by the "EQ-5D-5L" | 9 months after inclusion
  "EQ-5D-5L" index score and EQ-VAS score (range 0-100) where higher scores indicates better health-related quality of life.
Health-related quality of life assessed by the "EQ-5D-5L" | 15 months after inclusion
  "EQ-5D-5L" index score and EQ-VAS score (range 0-100) where higher scores indicates better health-related quality of life.
Health-related quality of life assessed by the "EQ-5D-5L" | 21 months after inclusion
  "EQ-5D-5L" index score and EQ-VAS score (range 0-100) where higher scores indicates better health-related quality of life.
Disease-specific quality of life assessed by "Amyotrophic lateral sclerosis assessment scale - 5 items (ALSAQ-5)" | At inclusion
  "ALSAQ-5" score (range 0-100), with 0 reflecting the best health state
Disease-specific quality of life assessed by "Amyotrophic lateral sclerosis assessment scale - 5 items (ALSAQ-5)" | 3 months after inclusion
  "ALSAQ-5" score (range 0-100), with 0 reflecting the best health state
Disease-specific quality of life assessed by "Amyotrophic lateral sclerosis assessment scale - 5 items (ALSAQ-5)" | 9 months after inclusion
  "ALSAQ-5" score (range 0-100), with 0 reflecting the best health state
Disease-specific quality of life assessed by "Amyotrophic lateral sclerosis assessment scale - 5 items (ALSAQ-5)" | 15 months after inclusion
  "ALSAQ-5" score (range 0-100), with 0 reflecting the best health state
Disease-specific quality of life assessed by "Amyotrophic lateral sclerosis assessment scale - 5 items (ALSAQ-5)" | 21 months after inclusion
  "ALSAQ-5" score (range 0-100), with 0 reflecting the best health state
Health-related quality of life assessed by "Severe Respiratory Insufficiency Questionnaire" | At inclusion
  "Severe Respiratory Insufficiency Questionnaire" score (range 0-100), with 100 reflecting the best health state.
Health-related quality of life assessed by "Severe Respiratory Insufficiency Questionnaire" | 3 months after inclusion
  "Severe Respiratory Insufficiency Questionnaire" score (range 0-100), with 100 reflecting the best health state.
Health-related quality of life assessed by "Severe Respiratory Insufficiency Questionnaire" | 9 months after inclusion
  "Severe Respiratory Insufficiency Questionnaire" score (range 0-100), with 100 reflecting the best health state.
Health-related quality of life assessed by "Severe Respiratory Insufficiency Questionnaire" | 15 months after inclusion
  "Severe Respiratory Insufficiency Questionnaire" score (range 0-100), with 100 reflecting the best health state.
Health-related quality of life assessed by "Severe Respiratory Insufficiency Questionnaire" | 21 months after inclusion
  "Severe Respiratory Insufficiency Questionnaire" score (range 0-100), with 100 reflecting the best health state.
Health-related quality of life assessed by "Kidsscreen-27" | At inclusion
  "Kidsscreen-27" score where mean (±SD) scores of 50 ± 10 define normality for children and adolescents aged 8-18 years across Europe. Higher scores indicate a better health-related quality of life.
Health-related quality of life assessed by "Kidsscreen-27" | 3 months after inclusion
  "Kidsscreen-27" score where mean (±SD) scores of 50 ± 10 define normality for children and adolescents aged 8-18 years across Europe. Higher scores indicate a better health-related quality of life.
Health-related quality of life assessed by "Kidsscreen-27" | 9 months after inclusion
  "Kidsscreen-27" score where mean (±SD) scores of 50 ± 10 define normality for children and adolescents aged 8-18 years across Europe. Higher scores indicate a better health-related quality of life.
Health-related quality of life assessed by "Kidsscreen-27" | 15 months after inclusion
  "Kidsscreen-27" score where mean (±SD) scores of 50 ± 10 define normality for children and adolescents aged 8-18 years across Europe. Higher scores indicate a better health-related quality of life.
Health-related quality of life assessed by "Kidsscreen-27" | 21 months after inclusion
  "Kidsscreen-27" score where mean (±SD) scores of 50 ± 10 define normality for children and adolescents aged 8-18 years across Europe. Higher scores indicate a better health-related quality of life.
Caregiver burden assessed by "Zarit Burden Interview" | At inclusion
  "Zarit Burden Interview" total score (range 0-88 where a higher score indicates greater burden).
Caregiver burden assessed by "Zarit Burden Interview" | 3 months after inclusion
  "Zarit Burden Interview" total score (range 0-88 where a higher score indicates greater burden).
Caregiver burden assessed by "Zarit Burden Interview" | 9 months after inclusion
  "Zarit Burden Interview" total score (range 0-88 where a higher score indicates greater burden).
Caregiver burden assessed by "Zarit Burden Interview" | 15 months after inclusion
  "Zarit Burden Interview" total score (range 0-88 where a higher score indicates greater burden).
Caregiver burden assessed by "Zarit Burden Interview" | 21 months after inclusion
  "Zarit Burden Interview" total score (range 0-88 where a higher score indicates greater burden).

CONTACTS AND LOCATIONS:
Overall Officials: Ole-Bjørn Tysnes, Principal Investigator — Haukeland University Hospital
Locations (9):
- Norway (9):
  - Nordland Hospital Bodø, Bodø, Nordland
  - Sørlandet Hospital Trust, Kristiansand, Vest Agder
  - Haukeland University Hospital, Bergen
  - Akershus University Hospital, Lørenskog
  - Oslo University Hospital, Oslo
  - Østfold Hospital Kalnes, Sarpsborg
  - Stavanger University Hospital, Stavanger
  - Universitetssykehuset Nord-Norge, Tromsø
  - St. Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No